CLINICAL TRIAL: NCT00417014
Title: Hodgkins Disease Study
Brief Title: Combination Chemotherapy and/or Radiation Therapy in Treating Young Patients With Hodgkin's Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CCLG-HD-8201; CDR0000454559 (Registry Identifier: PDQ (Physician Data Query)); EU-20585
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2006-12

CONDITIONS: Lymphoma
Keywords: stage I childhood Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage III childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — Chlorambucil; Prednisolone; Procarbazine; Vinblastine; Radiotherapy

INTERVENTIONS:
Drug: chlorambucil
Drug: prednisolone
Drug: procarbazine hydrochloride
Drug: vinblastine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as chlorambucil, vinblastine, procarbazine, and prednisolone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill cancer cells. Giving more than one drug (combination chemotherapy) together with radiation therapy may kill more cancer cells.

PURPOSE: This clinical trial is studying how well giving combination chemotherapy and/or radiation therapy works in treating young patients with Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Establish a uniform practice for the management of children with Hodgkin's lymphoma.
* Document the long-term side effects of such management.
* Establish whether or not children can be safely managed without staging laparotomy and splenectomy.
* Establish whether or not chlorambucil, vinblastine, procarbazine hydrochloride, and prednisolone (CLVPP) is an effective alternative to mechlorethamine, vincristine, procarbazine hydrochloride, and prednisone (MOPP) chemotherapy.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 3 treatment regimens according to disease stage and presence of bulky mediastinal disease.

* Involved-field radiotherapy (for patients with stage IA [nodal] disease): Patients undergo involved-field radiotherapy 5 days a week for 4 weeks.
* CLVPP chemotherapy (for patients with all other stages of disease AND no bulky mediastinal disease): Patients receive CLVPP chemotherapy comprising oral chlorambucil, oral procarbazine hydrochloride, and oral prednisolone on days 1-14 and vinblastine IV on days 1 and 8. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
* CLVPP chemotherapy and radiotherapy (for patients with all other stages of disease AND bulky mediastinal disease): Patients receive CLVPP chemotherapy as above. Patients then undergo radiotherapy to the mediastinum beginning 2 weeks after completing the last course of CLVPP chemotherapy.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 358 patients were accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Biopsy proven Hodgkin's lymphoma

  * Any stage allowed

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 358 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Martin, MD, Study Chair — Royal Liverpool Children's Hospital, Alder Hey; A. Barratt, MD — Royal Marsden NHS Foundation Trust